CLINICAL TRIAL: NCT04098380
Title: A Randomized Controlled Trial on Small Versus Large Bite Closure of Emergency Midline Laparotomy
Brief Title: Small Versus Large Bite Closure of Emergency Midline Laparotomy
Acronym: E-STITCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Mansoura104
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small bite (Active Comparator): The needle bites will be applied with a bite width of 5 mm and inter-suture spacing of 5 mm
  Interventions: Procedure: Small Bite
- Large bite (Active Comparator): The needle bites will be applied with a width of 10 mm and inter-suture spacing of 10 mm
  Interventions: Procedure: Larger bite

INTERVENTIONS:
Procedure: Small Bite — the bites will be applied with a bite width of 5 mm and inter-suture spacing of 5 mm
  Arms: Small bite
Procedure: Larger bite — the bites will be applied with a width of 10 mm and inter-suture spacing of 10 mm
  Arms: Large bite

SUMMARY:
In daily practice, midline laparotomy is an incision frequently performed by surgeons to achieve a rapid and wide access to the abdomen. However, incisional hernia stands as the most common complication following this type of incision, with an incidence reaching up to 20% and even higher in the case of emergency laparotomy.

A recent randomized controlled trial compared small bite sutures and large bite closure of elective midline laparotomy and reported a significant decrease of incisional hernia rate from 18% to 5.6% in favor of small-bite technique. These promising results were subsequently confirmed in a wide-scale multicenter double-blinded randomized trial, the STITCH study.

The investigators will conduct this randomized controlled trial to compare the small tissue bite (SB) technique and the large bite (LB) technique for closure of emergency midline laparotomy. The main outcome of the study will be the incidence of incisional hernia within one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes aging less than 70 years old

Exclusion Criteria:

* All procedures which will be performed on elective basis will be excluded
* patients who are pregnant.
* Patients on systemic steroid or chemotherapy
* patients with incisional hernia or fascial defect; and/or relaparotomy within 30-days of another surgical intervention.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-09-21 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 12 months after surgery
  Diagnosis of incisional hernia within 12 months after surgery by clinical examination or by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No